CLINICAL TRIAL: NCT03771833
Title: Comparison of M5 and M6 Versions of the MARIA Imaging System on Patients Attending Symptomatic Breast Clinic in Cheltenham, United Kingdom (UK), Including a Sub-study to Research the Dielectric Constant of Aspirated Cyst Fluid
Brief Title: M5 vs. M6 Comparison Study With a Sub Study Into the Dielectric Constant of Aspirated Cyst Fluid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Micrima, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PROT-P2-024
Record Dates: First submitted 2018-11-29; First posted 2018-12-11 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Breast Cyst; Breast Cancer Female
Keywords: breast; cancer; breast cancer; imaging
MeSH Terms: conditions — Breast Cyst; Neoplasms; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Main MARIA scan visit (Other): For Arm 1, participants will be identified in clinic as having a suitable symptomatic breast and approached about the study. They will have the study design explained to them and will be informed that they are under no obligation to participate. Arm 1 participants will receive study information that they will be sent home with and informed that they will be approached via a telephone call in 2-3 days (or the closest working day to that date) to enquire if they would like to schedule an appointment for the study visit. If so, this will be scheduled to occur around 7 days from the date of the phone call.
  Interventions: Device: MARIA scan
- Same-day MARIA scan visit (Other): For Arm 2, participants will be identified in clinic as having a suitable symptomatic breast and approached about the study. They will have the study design explained to them and will be informed that they are under no obligation to participate. Arm 2 participants will receive study information and as much time as possible to consider their involvement with the study (at least 1 hour). If the patient agrees to participate, they will be scheduled to have their MARIA scans at a time that suits their commitments that day.
  This arm also includes the 2b group, who can optionally consent to a dielectric constant reading of their routinely-aspirated cyst fluid before this is disposed of as per usual site process.
  Interventions: Device: MARIA scan

INTERVENTIONS:
Device: MARIA scan — The MARIA breast imaging system comprises of a scanning unit, housed under a patient bed. The scanning unit houses a hemispherical array, into which varying sizes of insert are fitted to ensure a close fit to the breast. The patient lies prone on the bed with their breast pendulous through an aperture in the bed and the scanning unit is risen to meet the breast. The fit is non-compressing and the scanner does not use ionising radiation.

SUMMARY:
The MARIA breast imaging system is a Conformité Européenne (CE)-marked radio-frequency (RF) medical imaging device. The system employs an electromagnetic imaging technique that exploits the dielectric contrast between normal and cancerous tissues. The performance and imaging characteristic differences between the M5 and M6 versions of MARIA are not yet well demonstrated in the clinical environment, particularly with regards to cysts. The evaluation of some aspects of this potentially important new technology will occur in this comparative technical study. Further, the dielectric constant of cyst fluid is currently not well understood and obtaining readings from aspirated cyst fluid in applicable patients will be attempted.

ELIGIBILITY:
Inclusion Criteria:

* attending a symptomatic breast care clinic at the study site
* have a palpable lump in the breast
* female sex
* 18 years or older
* able to provide informed consent
* not in any identified vulnerable group

Exclusion Criteria:

* unable to mount MARIA patient bed using provided 2-step
* unable to lie in the prone position for a period of up to 15 minutes
* patient who have undergone biopsy less than 5 days before the MARIA scan
* patient with implanted electronics
* patient with breast implants
* patients with nipple piercings (unless they are removed prior to the MARIA scan)
* breast size too small or too large to be suitable for both arrays

Further:

* participants with a large cyst or cysts that require draining at their clinical appointment will not be eligible for Arm 1, as the procedure to drain their cyst will change the appearance of the cyst from the imaging that they have done that day to the MARIA image obtained around 10 days later
* Arm 1 and 2 are mutually exclusive

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The device is currently registered for the scanning of female human breast tissue only
Enrollment: 22 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Establish the presence or absence of a difference in the MARIA(R) outputs obtained with M5 and M6 when the participants is not moved between scans and when they are moved between scans | Up to 12 weeks
  This will be established from Arm 1 and Arm 2 by scanning the participant between both versions of the MARIA system. As has been investigated in-house with healthy volunteers, the patient will take part in a series of scans that will involve them remaining stationary between scans, and moving between scans. The differences between these images will be analysed, using the known palpable lesion in the breast as a landmark.
Establish the presence or absence of a difference between MARIA(R) outputs on the same device when the participant is stationary between scans and when they are moved between scans | Up to 12 weeks
  This will be established from Arm 1 and Arm 2 by scanning the participant on each separate version of the MARIA system. As has been investigated in-house with healthy volunteers, the patient will take part in a series of scans that will involve them remaining stationary between scans, and moving between scans. The differences between these images will be analysed, using the known palpable lesion in the breast as a landmark.
Measure the dielectric constant of aspirated cyst fluid and any variance between cyst type | Up to 12 weeks
  This will be established from Arm 2b by recording the dielectric constant of the aspirated cyst fluid as soon as possible after aspiration using a dielectric probe. No cysts will be aspirated exclusively for this procedure and fluid will be disposed of as per usual site practice once the recording has taken place. Each cyst fluid sample will have its dielectric constant recorded three times and recorded in the provided software before disposal.

SECONDARY OUTCOMES:
Assess the diagnostic accuracy of both the M5 and M6 versions of the MARIA system in identifying lesions of the breast, including benign lesions such as cysts | Up to 12 weeks
  This will be established from Arm 1 and 2 by using a combination of reader results from clinician reads performed by the site team with all available clinical information and blind reads performed in house which will utilise no clinical information.
Understand participant acceptability of the MARIA scan and obtain feedback on patient experience: questionnaire | Up to 12 weeks
  This will be established from Arm 1 and 2 by asking the participant to complete a questionnaire of their experience after their participation in either of the two main study arms. The questionnaire comprises of 8 questions and a free-text box for any additional comments. The first two questions ask a participant to pick one of 5 options, from very easy to very difficult or very comfortable to very uncomfortable. The next even questions are Yes or No questions, with options for the participant to answer these as "Not sure" or "Not applicable" as appropriate. The questionnaire then ends with a free-text box for feedback.

CONTACTS AND LOCATIONS:
Locations (1):
- Thirlestaine Breast Centre, Gloucestershire Hospitals NHS Foundation Trust, Cheltenham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data collected will be anonymised